CLINICAL TRIAL: NCT02265601
Title: End-of-Life Health Care Decisions by Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Michael J. Green, Professor of Humanities, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RSGHP-08-005-01-CPHPS; RSGHP-08-005-01-CPHPS (Other Grant/Funding Number: ACS)
Record Dates: First submitted 2014-07-30; First posted 2014-10-16 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Neoplasms
Keywords: advance care planning; living wills; end of life; cancer
MeSH Terms: conditions — Neoplasms; Death | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- computer-based decision aid (Experimental): "Making Your Wishes Known: Planning Your Medical Future"- Offers tailored education, values clarification exercises, and a sophisticated decision aid that translates an individual's goals and preferences into a specific medical plan that can be implemented by a health care team.
  Interventions: Other: computer-based decision aid
- standard care (Active Comparator): paper/pencil living will form
  Interventions: Other: standard care

INTERVENTIONS:
Other: computer-based decision aid — Offers tailored education, values clarification exercises, and a sophisticated decision aid that translates an individual's goals and preferences into a specific medical plan that can be implemented by a health care team.
  Other Names: "Making Your Wishes Known: Planning Your Medical Future"
  Arms: computer-based decision aid
Other: standard care — paper/pencil living will form
  Arms: standard care

SUMMARY:
This study is designed to help the investigators understand more about how people plan for their future medical needs, a process known as "advance care planning."

The study is under the direction of Michael J. Green, M.D., and Benjamin Levi, M.D. physicians at Penn State Hershey Medical Center.

Participation in the project takes place during a single visit to the Medical Center campus. During this one-to-three hour visit, participants complete several questionnaires and use a computer program that produces a printed advance directive that can be shared with their physicians and loved ones. Participants will receive compensation toward travel expenses.

DETAILED DESCRIPTION:
Background: Despite widespread agreement that individuals ought to plan for their medical futures, few people (even seriously ill patients with cancer) actually complete advance directives, fewer yet understand key elements, and even when advance directives do exist, there are often barriers to their being implemented.

Objectives: The investigators innovative, multimedia, interactive, computer-based decision aid, "Making Your Wishes Known: Planning Your Medical Future," offers tailored education, values clarification exercises, and a sophisticated decision aid that translates an individual's goals and preferences into a specific medical plan that can be implemented by a health care team. This project aims to evaluate its impact on decision-making and health care received by individuals at the end of life in a randomized clinical trial among a population of patients with advanced cancer who have life expectancies of < 12 months.

Specific Aims:

Aim 1: To evaluate the impact of a computer-based advance care planning intervention on end-of-life decision-making by cancer patients with estimated life expectancies < 12 months. The investigators hypothesize that, compared to standard care (paper/pencil living will form), use of the computer-based intervention will:

H1: Improve individuals' decision-making about end-of-life health care

H2: Improve individuals' experience with the process of advance care planning

H3: Not increase individuals' hopelessness or anxiety, nor harm the doctor-patient relationship

Aim 2: To evaluate the impact of the investigators intervention on end-of-life health care received by cancer patients with estimated life expectancies < 12 months. The investigators hypothesize that, compared to standard care, use of the computer intervention will:

H4: Increase physician awareness of individuals' health care wishes

H5: Increase physician adherence to individuals' health care wishes

Study Design: Randomized, controlled pre-intervention/post-intervention trial comparing a computer-based educational intervention with standard care

Cancer Relevance: Patients with advanced cancer face many medical decisions, some of which must be made when the patient cannot speak for him or herself. Helping these individuals to effectively articulate and communicate their wishes, in advance, can help assure that treatment they receive is consistent with their values, goals and wishes. This study aims to test the effectiveness of the investigators' computer-based intervention. If successful, this intervention can help improve the quality of health care received by cancer patients at the end of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to give informed consent
* interested in participating in advance care planning
* able to read and understand English at an 8th grade level (per WRAT-3 screening test)
* advanced cancer (primary or metastatic), with estimated lifespan < 6 months (as determined by their treating physician)
* cognitively able to engage in advance care planning (Mini Mental State Exam (MMSE) score >23)
* absence of moderate or severe depression (BDI-II score <20/63)

Exclusion Criteria:

* unable to read and understand English at an 8th grade level (per Wide Range Achievement Test (WRAT-3))
* not cognitively able to engage in advance care planning (Mini Mental State Exam (MMSE) score < 23)
* moderate or severe depression (BDI-II score >20/63)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Participant knowledge of advance care planning | Pre and post-intervention
  Knowledge of advance care planning will be compared between control and intervention groups, using a true/false and multiple choice questionnaire about advance care planning.

SECONDARY OUTCOMES:
Participant decisional conflict | post-intervention
  Assessment of conflict associated with making end-of-life decisions will be assessed with the decisional conflict scale.
Participant satisfaction with decision | post-intervention
  Assessment of satisfaction with decisions associated with advance care planning will be assessed with the satisfaction with decision scale.
Participant satisfaction with advance care planning | post-intervention
  Satisfaction with with advance care planning process will be compared between intervention and control group with a satisfaction questionnaire.
Participant self-determination | pre and post-intervention
  Self determination will be compared between intervention and control group with a self-determination questionnaire.
Participant anxiety | pre and post-intervention
  Pre and post-intervention anxiety will be compared between intervention and control group with the state trait anxiety instrument.
Participant hopelessness | pre and post-intervention
  Assessment of pre and post-intervention hopelessness will be compared between intervention and control group using the Beck Hopelessness scale and a measure of hopefulness.
Physician awareness of patients' health care wishes | post-death chart review
  Comparison will be made between intervention and control group regarding whether an advance directive is present in the patient's medical record, and whether the physician is aware of the patient's wishes.
Physician adherence to patients' health care wishes | post-death chart review
  Comparison will be made between intervention and control group regarding whether patients' wishes are followed at the end of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Green, MD, MS, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center